CLINICAL TRIAL: NCT04236011
Title: Exploratory Study to Evaluate Efficacy and Safety of GC012F Injection in BCMA+ Refractory/Relapsed Multiple Myeloma
Brief Title: BCMA and CD19 Targeted Fast Dual CAR-T for BCMA+ Refractory/Relapsed Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Weijun Fu, Director of Hematology Department, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBF002
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Multiple Myeloma
Keywords: Fast; Chimeric Antigen Receptor T; BCMA; CD19; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Fasting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC012F treatment (Experimental): BCMA+ R/R multiple myeloma patients be treated with a single dose of GC012F cells. Total dose of (1-5)*10E5/kg cells will be administered at Day 0.
  Interventions: Biological: GC012F injection

INTERVENTIONS:
Biological: GC012F injection — GC012F injection is a autologous dual CAR-T targeted BCMA and CD19. A single infusion of CART cells will be administered intravenously.

SUMMARY:
This is a single arm, open-label, multi-center prospective study to determine the safety and efficacy of GC012F CAR-T cells in patients diagnosed with BCMA+ refractory/relapsed multiple myeloma (r/r MM).

DETAILED DESCRIPTION:
The main aim of the study is to determine the safety and efficacy of GC012F in r/r MM. GC012F is an autologous dual chimeric antigen receptor T-cell (CAR-T) therapy that targets B-cell maturation antigen (BCMA) and CD19. This study comprises of a Screening Phase (less than or equal to [<=] 28 days prior to apheresis) followed by Apheresis (will occur upon enrollment); Treatment Phase including a conditioning regimen followed by infusion of GC012F and post-infusion assessments from Day 1 to Day 84; and a Post-treatment Phase (Day 85 and up to end of the study). Efficacy will be explored to assessed and safety will be closely monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed prior diagnosis of active multiple myeloma as defined by the updated IMWG criteria;
2. Diagnosis of MM with relapsed or refractory disease. Definition of Refractory/relapse:

   1. Have had at least 3 prior lines of therapy or primary refractory as defined by Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Prior therapy should include PI and IMiD. Note: Patients should undergone at least have at least complete 1 cycle treatment in each line. Induction with or without hematopoietic stem cell transplant followed by maintenance therapy is considered a single line of therapy.
   2. Have had at least 2 prior lines of therapy when refractory to both immunomodulatory drug (IMiD) and proteasome inhibitor(PI) (Refractory was defined by IMWG consensus criteria);
3. Estimated life expectancy ≥3 months;
4. Hemoglobin ≥ 8.0 g/dL;
5. Absolute neutrophil count ≥ 0.75*10E9/L;
6. Platelet count ≥ 50*10E9/L;
7. Absolute lymphocyte count ≥ 1*10E8/L;
8. Liver, kidney and cardiopulmonary functions meet the following requirements: a)Total bilirubin ≤ 2×ULN(except for Gilbert Syndrome); ALT and/or AST ≤3 × ULN; b)clearance of serum creatinine ≥ 40 mL/min, calculated by Cockcroft-Gault; c)Corrected serum calcium ≤ 12.5mg/dL or free ion calcium ≤ 6.5mg/dL(1.6mmol/L);
9. Sufficient venous access for leukapheresis collection, and no other contraindications to leukapheresis;
10. Subjects and sexual partner with fertility are willing to use effective and reliable method of contraception for at least 100 days after CART cell infusion;
11. Subjects must have signed written, informed consent.

Exclusion Criteria:

1. Accompanied by other uncontrolled malignancies.There are two exceptions to this criterion: Recepted radical therapy carcinoma without activity within 3 years before screening; and fully treated skin non-melanoma;
2. Any situations not benefit for subjects to accept or tolerated to planned therapy or understand informed consent; or any situation in which investigators believe that participation in this study is not in the subject's best interests (e.g., harm to health), or any situation that may prevent, limit or confuse the assessment;
3. Convulsion or stoke within past 6 months;
4. Any instability of systemic disease within 6 months prior to screening, including but not limited to congestive heart failure (New York heart association (NYHA) classification ≥ III), unstable angina, cerebrovascular accident, or transient cerebral ischemic, myocardial infarction,LEVF< 45% (assessed by an echocardiogram or multi-door circuit scan );
5. Patients have central nervous system (CNS) metastases or CNS involvement (including cranial neuropathies or mass lesions and leptomeningeal disease);
6. Subjects with positive HBsAg or HBcAb postive and peripheral blood HBV DNA titer is higher than the lower limit of detection of the research institution; HCV antibody positive; HIV antibody positive; syphilis primary screening antibody positive;
7. Presence or suspicion of fungi, bacteria, viruses or other infections that are uncontrollable or requiring intravenous treatment;
8. Activity of autoimmune diseases (such as crohn's disease, rheumatoid arthritis, systemic lupus erythematosus), orhistory of autoimmune disease within the last 3 years;
9. Clinical evidence of dementia or changes of mental state.
10. Exist of pulmonary fibrosis;
11. Allergy subjects or history of severe hypersensitivity;
12. Oxygen inhalation requirment to maintain adequate oxygen saturation;
13. Surgery (except for local anesthesia surgery) plan 2 weeks before apheresis. during or 2 weeks after CART infusion;
14. Chemotherapy forbidden for cyclophosphamide or fludarabine;
15. Pregnant or lactating, or planning to have a pregnancy during or within 100 days after treatment;
16. Patients who are accounted to be not appropriate for this trail by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events after GC012F infusion | up to 24 weeks after GC012F infusion

SECONDARY OUTCOMES:
Percentage of MRD negative patients after GC012F treatment | 12 weeks, 24 weeks after GC012F infusion
ORR (PR, VGPR, CR and sCR) of patients receive GC012F treatment | 12 weeks, 24 weeks after GC012F infusion
Progression free survival after GC012F treatment | 12 weeks, 24 weeks after GC012F infusion
Copies and cell counts of CAR in blood and bone marrow (if available) after GC012F treatment | Days 4, 7, 10, 14 and weeks 4, 8, 12, 18, 24 after GC012F infusion
  Bone marrows will be collected in weeks 4, 8, 12, 18, 24 after GC012F infusion.
Cytokines in serum after GC012F treatment | Days 4, 7, 10, 14 and weeks 4, 8, 12, 18, 24 after GC012F infusion
Subset of lymphocytes and ADA in blood after GC012F treatment | Weeks 4, 8, 12, 18, 24 after GC012F infusion
Replication competent lentivirus (RCL) in blood after GC012F treatment | Weeks 4, 12, 24 after GC012F infusion
Duration of response after GC012F treatment | 12 weeks, 24 weeks after GC012F infusion
Overall survival after GC012F treatment | 12 weeks, 24 weeks after GC012F infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided